CLINICAL TRIAL: NCT06953687
Title: Implementing and Evaluating a Patient-Centered PTSD Treatment Program for Military Personnel
Brief Title: Shared Decision Making in PTSD Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Vanessa Jacoby, Associate Professor, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00001302; HT9425-23-2-0016 (Other Grant/Funding Number: Department of Defense); HT94252320018 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2025-04-22; First posted 2025-05-01 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Post Traumatic Stress Disorder PTSD
Keywords: Shared Decision Making; Patient Characteristics; Patient Treatment preference; Treatment engagement; Treatment outcomes
MeSH Terms: conditions — Combat Disorders | interventions — 2-cyclohexylidenhydrazo-4-phenyl-thiazole

STUDY DESIGN:
Intervention Model Description: Two-stage randomized preference design to examine relationship between patient characteristics, treatment preferences and treatment outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Prolonged Exposure (PE) Therapy Massed (Experimental): Daily treatment sessions Monday-Friday for up to 24 sessions
  Interventions: Behavioral: Prolonged Exposure Therapy; Other: Shared Decision Making (SHARE)
- Prolonged Exposure (PE) Spaced (Experimental): Weekly treatment formula for up to 24 sessions
  Interventions: Behavioral: Prolonged Exposure Therapy; Other: Shared Decision Making (SHARE)
- Cognitive Processing Therapy (CPT) Massed (Experimental): Daily treatment sessions Monday-Friday for up to 24 sessions
  Interventions: Behavioral: Cognitive Processing Therapy; Other: Shared Decision Making (SHARE)
- Cognitive Processing Therapy (CPT) spaced (Experimental): Weekly treatment formula for up to 24 sessions
  Interventions: Behavioral: Cognitive Processing Therapy; Other: Shared Decision Making (SHARE)
- Written Exposure Therapy (WET) Massed (Experimental): Daily treatment sessions Monday-Friday for up to 24 sessions
  Interventions: Behavioral: Written Exposure Therapy; Other: Shared Decision Making (SHARE)
- Written Exposure Therapy (WET) Spaced (Experimental): Weekly treatment formula for up to 24 sessions
  Interventions: Behavioral: Written Exposure Therapy; Other: Shared Decision Making (SHARE)

INTERVENTIONS:
Behavioral: Prolonged Exposure Therapy — PE is a cognitive-behavioral treatment for PTSD that is typically delivered in ten 90-minute sessions . For the current study using a variable length approach, participants may complete up to 24 sessions. Based on emotional processing theory PE addresses trauma-related avoidance of thoughts, behaviors, and situations, as well as unhelpful beliefs about oneself, others, and the world that were learned as a result of trauma.
  Other Names: PE
  Arms: Prolonged Exposure (PE) Spaced; Prolonged Exposure (PE) Therapy Massed
Behavioral: Cognitive Processing Therapy — CPT is a 12-session, cognitive behavioral PTSD treatment typically delivered in 60-minute sessions that can be personalized to include fewer or additional sessions. For the current study using a variable length approach, participants may complete up to 24 sessions. CPT is based in cognitive theory and posits that impeded recovery following trauma occurs due to unhelpful and unrealistic beliefs that may develop after trauma, leading to chronic anger, guilt, shame, and avoidance of trauma reminders. During CPT, patients learn about PTSD symptoms, impeded recovery and cognitive theory, and the connection between trauma-based thoughts and feelings.
  Other Names: CPT
  Arms: Cognitive Processing Therapy (CPT) Massed; Cognitive Processing Therapy (CPT) spaced
Behavioral: Written Exposure Therapy — WET is a cognitive behavioral therapy for PTSD that typically consists of 5 weekly 50-minute sessions. For the current study using a variable length approach, participants may complete up to 7 sessions. WET is based on an extinction and emotional processing treatment model. First, patients learn about PTSD and the role of avoidance in maintaining PTSD symptoms. Next, patients are guided to write about their trauma for 30 minutes and afterwards, the therapist briefly checks in with the patient. This procedure is followed for the next 4 sessions, with guidance to first write about the trauma, and in later sessions to write about consequences of the trauma and the patient's current meaning of their lives. The goals of WET are to assist the patient in emotionally processing the event and reduce avoidance of trauma-related thoughts and memories, which facilities recovery.
  Other Names: WET
  Arms: Written Exposure Therapy (WET) Massed; Written Exposure Therapy (WET) Spaced
Other: Shared Decision Making (SHARE) — The study will use the SHARE Approach to facilitate treatment planning and decision-making. SHARE stands for:
  1. Seek the patient's participation
  2. Help the patient explore and compare treatment options
  3. Assess the patient's values and preferences
  4. Reach a decision with the patient
  5. Evaluate the patient's decision The Shared Decision Making Patient Preference Checklist will be used to determine the participant's preference for type of treatment, frequency of treatment sessions, and treatment delivery modality. Step 5 also includes following up with the patient and making changes if something it not working well for the patient.
  Other Names: SHARE

SUMMARY:
The purpose of this research study is to learn about how Shared Decision Making, when used to decide treatment, impacts treatment engagement, retention, and outcomes for active duty military personnel seeking treatment for posttraumatic stress disorder (PTSD).

Shared Decision Making between the service member and the therapists will be used to match patients to 1 of 3 different types of therapy for PTSD: (1) Prolonged Exposure (PE) therapy, (2) Cognitive Processing Therapy (CPT), or (3) Written Exposure Therapy (WET) in 1 of 2 different frequencies: (1) massed (daily) or (2) spaced (weekly).

DETAILED DESCRIPTION:
The primary objectives of the project are to evaluate the relationships between patient characteristics, patient treatment preferences, treatment engagement, and treatment outcomes for active duty services members engaging in a Shared Decision Making pre-intervention followed by evidence-based PTSD treatment. A secondary objective is to evaluate the impact of Shared Decision Making to match patients to evidence-based cognitive behavioral treatments for PTSD.

Aim 1: To conduct a partially randomized preference trial to examine the relationships between patient characteristics, treatment preferences, and treatment outcomes for active duty service members engaging in a Shared Decision Making pre-intervention followed by evidence-based treatment for PTSD.

Research Question 1: What are the PTSD treatment initiation rates and completion rates for active duty service members engaging in a Shared Decision Making pre-intervention prior to starting an evidence-based treatment for PTSD?

Research Question 2: Will patient characteristics (i.e., age, gender, military pay grade, racial-ethnic identity, deployment history) predict patient preference for a treatment type, session frequency, or treatment modality?

Research Question 3: Will strength of preference in a specific treatment type, session frequency, or treatment modality predict PTSD treatment initiation, treatment completion, or PTSD symptom reduction?

Aim 2: To evaluate the impact of Shared Decision Making on PTSD treatment completion and PTSD symptom reduction for active duty military personnel.

Hypothesis 1: Patients who engage in Shared Decision Making will show higher rates of treatment completion as compared to prior PTSD randomized controlled trials (RCTs) with active duty service members

Hypothesis 2: Patients who engage in Shared Decision Making will show larger reductions in PTSD symptoms from pre-to posttreatment as compared to benchmarked outcomes from prior PTSD RCTs with active duty service members. Treatment gains will be maintained over time, consistent with prior research.

ELIGIBILITY:
Inclusion Criteria:

1. Adult active duty military service members aged 18 or older.
2. Meets diagnostic criteria for PTSD based on the Clinician Administered PTSD Scale for the Diagnostic and Statistical Manual of Mental Disorders-5 (CAPS-5).

Exclusion Criteria:

1. Acute suicidality or homicidality requiring immediate intervention, such as hospitalization.
2. Moderate to severe brain injury as assessed by the History of Head Injury Form
3. Severe alcohol consumption patterns as assessed using the Alcohol Use Disorders Identification Test and warranting immediate intervention as determined by clinical judgement.
4. Experiencing active psychosis or mania as determined by scores on the Prodromal Questionnaire and Mood Disorder Questionnaire in combination with clinical judgement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-05-09 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Completion of treatment initiation | Baseline to Treatment Session 1 (approximately 2 weeks)
  Percentage of participants initiate and complete at least one session of evidence-based Posttraumatic Stress Disorder (PTSD) treatment
Completion of all Treatment sessions | Baseline to Posttreatment (between 2 months and 7 months, depending on treatment selected and speed of progress)
  The percentage of participants who complete all manualized protocol sessions (i.e., 10 PE sessions, 12 CPT sessions, or 5 WET sessions) or (2) complete treatment early because they have achieved their treatment goals. This will be defined as achieving a 10 point reduction in on the PCL-5 and scoring below the diagnostic cutoff (a PCL- 5 score of ≤ 30), as well as the therapist and patient agreeing that treatment relevant goals have been met.
Preference for type of treatment | Measured at Pre-Treatment Shared Decision-Making Session
  Measured on a Likert Scale from 0= no preference to 10= extremely high preference
Posttraumatic Stress Disorder Checklist (PCL-5) | Baseline to 1 month follow up assessment (between 2 months and 7 months, depending on treatment selected and speed of progress)
  The PCL-5 is a 20-item self-report measure, selected for its dimensional sensitivity, with higher scores reflecting greater PTSD severity. Scoring is based on how much the patient has been bothered by the symptoms in the past month on a scale from "0 = not at all" to "4 = extremely. Scores range from 0-80 with a higher score indicating more severe PTSD.

SECONDARY OUTCOMES:
Brief Inventory of Psycho-social Functioning | Baseline to 1 month follow up assessment (between 2 months and 7 months, depending on treatment selected and speed of progress)
  7-item self-report instrument measuring respondents' level of functioning in seven life domains: romantic relationship, relationship with children, family relationships, friendships and socializing, work, training and education, and activities of daily living. Respondents indicate the degree to which they had trouble in the last 30 days in each area on a 7-point scale ranging from 0 ("Not at all") to 6 ("Very much"). Scores range from 0-42 with a higher score indicating better level of psycho-social function.
Patient Health Questionnaire 9 (PHQ-9) | Baseline to 1 month follow up assessment (between 2 months and 7 months, depending on treatment selected and speed of progress)
  9 items that assess both affective and somatic symptoms related to depression and depressive disorders; these 9 items correspond to the diagnostic criteria for Major Depressive Disorder. Respondents rate the frequency with which they have been bothered by depressive symptoms within the past two weeks on a scale ranging from 0 ("not at all") to 3 ("nearly every day"). Scores on all items are summed to obtain a total severity score between 0-27. Scores reflect no significant depressive symptoms (0-4), mild depressive symptoms (5-9), moderate depressive symptoms (10-14), moderately severe depressive symptoms (15-19), and severe depressive symptoms (>19)
Generalized Anxiety Disorder 7 (GAD-7) | Baseline to 1 month follow up assessment (between 2 months and 7 months, depending on treatment selected and speed of progress)
  This is a 7-item measure that asks participants to rate the frequency with which they have been bothered by anxiety symptoms within the past two weeks on a scale ranging from 0 ("not at all") to 3 ("nearly every day"). Scores on all items are summed to obtain a total severity score between 0-21. Scores reflect no significant anxiety symptoms (0-4), mild anxiety symptoms (5-9), moderate anxiety symptoms (10-14), and severe anxiety symptoms (>15).
Depressive Symptom Index - Suicidality Subscale (DSI-SS) | Baseline to 1 month follow up assessment (between 2 months and 7 months, depending on treatment selected and speed of progress)
  The DSI-SS is a 4-item self-report measure of suicidal ideation that focuses on ideation, plans, perceived control over ideation, and impulses for suicide occurring within the past two weeks. Scores on each item range from 0 to 3, with a total possible score from 0-12 with higher scores reflecting greater severity of suicidal ideation.
Posttraumatic Cognitions Inventory (PTCI) | Baseline to 1 month follow up assessment (between 2 months and 7 months, depending on treatment selected and speed of progress)
  The PTCI is a 36-item ( rated on a 7-point scale: 1=totally disagree and 7=totally agree) questionnaire that was developed to determine how an individual views the trauma and its sequelae in an attempt to understand both how PTSD develops and is maintained It is comprised of three subscales (Negative Cognitions about the Self (Score range 21-147), Negative Cognitions about the World (Score range 7-49), and Self-Blame (Score range 5-35)).
  Items 13, 32 and 34 are experimental, so not included in the subscales)
  Each subscale score is summed and then divided by the number of items to provide an average. The 3 subscale averages are totaled to give a total score between 33-221. A higher score indicates greater endorsement of negative conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Jacoby, PhD, Principal Investigator — The University of Texas Health Science Center at San Antonio; Alan L Peterson, PhD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (2):
- United States (2):
  - Carl R. Darnall Army Medical Center (CRDAMC), Fort Cavazos, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
As a STRONG STAR study, presentations and publications produced as a result of this work will follow the STRONG STAR Standard Operating Procedure STRONG STAR-ADM-001-5.0. The investigators will share deidentified date with other researchers.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: At completion of the study, summary results will be posted to ClinicalTrials.gov and after review and publication in a peer review journal.

REFERENCES:
- [Background] Resick PA, Wachen JS, Dondanville KA, LoSavio ST, Young-McCaughan S, Yarvis JS, Pruiksma KE, Blankenship A, Jacoby V, Peterson AL, Mintz J; STRONG STAR Consortium. Variable-length Cognitive Processing Therapy for posttraumatic stress disorder in active duty military: Outcomes and predictors. Behav Res Ther. 2021 Jun;141:103846. doi: 10.1016/j.brat.2021.103846. Epub 2021 Mar 25. PMID 33894644
- [Background] Foa EB, McLean CP, Zang Y, Rosenfield D, Yadin E, Yarvis JS, Mintz J, Young-McCaughan S, Borah EV, Dondanville KA, Fina BA, Hall-Clark BN, Lichner T, Litz BT, Roache J, Wright EC, Peterson AL; STRONG STAR Consortium. Effect of Prolonged Exposure Therapy Delivered Over 2 Weeks vs 8 Weeks vs Present-Centered Therapy on PTSD Symptom Severity in Military Personnel: A Randomized Clinical Trial. JAMA. 2018 Jan 23;319(4):354-364. doi: 10.1001/jama.2017.21242. PMID 29362795
- [Background] Sloan DM, Marx BP, Resick PA, Young-McCaughan S, Dondanville KA, Straud CL, Mintz J, Litz BT, Peterson AL; STRONG STAR Consortium. Effect of Written Exposure Therapy vs Cognitive Processing Therapy on Increasing Treatment Efficiency Among Military Service Members With Posttraumatic Stress Disorder: A Randomized Noninferiority Trial. JAMA Netw Open. 2022 Jan 4;5(1):e2140911. doi: 10.1001/jamanetworkopen.2021.40911. PMID 35015065